CLINICAL TRIAL: NCT00742300
Title: Phase I/II Open-Label Monocentric Clinical Trial for Induction of Tolerance With CD34-Enriched Autologous Hematopoietic Stem Cell Transplantation After High-Dose Chemotherapy With Cyclophosphamide and Rabbit-Antithymocyte Globulin for Refractory Autoimmune Diseases
Brief Title: Autologous Hematopoietic Stem Cell Transplantation for Refractory Autoimmune Diseases
Acronym: ASTRAD
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Christoph Krukenkamp, Charité Universitätsmedizin Berlin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-0198
Record Dates: First submitted 2008-08-26; First posted 2008-08-27 (Estimated); Last update posted 2008-11-24 (Estimated); Status verified 2008-11

CONDITIONS: Autoimmune Diseases
Keywords: ASCT; Tolerance induction; SLE; Transplantation; Autoimmune diseases
MeSH Terms: conditions — Autoimmune Diseases | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Treatment Group
  Interventions: Procedure: Autologous hematopoietic stem cell transplantation

INTERVENTIONS:
Procedure: Autologous hematopoietic stem cell transplantation — Transplantation of CD34-selected autologous hematopoietic stem cells after high-dose chemotherapy with cyclophosphamide (200mg/kg) and rabbit-antithymocyteglobulin (90mg/kg)
  Other Names: Mobilization: 2.0 g/m2 Cyclophosphamide followed by daily G-CSF (10 µg/kg, Amgen, Thousand Oaks, CA); Conditioning: 200mg/kg Cyclophosphamide (Endoxan), 90mg/kg rabbit-antithymocyteglobulin (ATG, Fresenius, Bad Homburg, Germany); Stem cell selection: CliniMACS Device (Miltenyi Biotec, Bergisch Gladbach, Germany)

SUMMARY:
While glucocorticoids and immunosuppressants ameliorate manifestations of autoimmune diseases in many patients, current therapies are insufficient to control the disease in a subset of patients, and their clinical prognosis remains poor due to the development of vital organ failure, cumulative drug toxicity and to the increased risk of cardiovascular disease and malignancy. Immunoablative chemotherapy followed by autologous hematopoietic stem cell transplantation (ASCT) has recently emerged as a promising experimental therapy for severely affected patients, providing them the potential to achieve treatment-free, long-term remission. The rationale for applying ASCT to autoimmune diseases has been the hope that immunoablation could eliminate inflammation-driving pathogenic cells from the immune system, and that regeneration of the patients' immune system from hematopoietic precursors could re-establish immunological tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Autoimmune disease
* Active disease with inadequate response to standard protocols (glucocorticoids and at least two different regimens of immunosuppressive drugs, such as intravenous cyclophosphamide 800-1000mg/application)
* Provision of informed consent by subject

Exclusion Criteria:

* Active or chronic infections
* Uncontrolled arrhythmia or congestive heart failure (ejection fraction below 50% determined by echocardiogram)
* Lung fibrosis (transfer factor for carbon monoxide [TLCO] <45%)
* renal insufficiency (glomerular filtration rate below 40 ml/min)
* Pulmonary arterial hypertension (>40mmHg)
* History of malignancy
* Women who are pregnant or breastfeeding
* Use non-reliable methods of contraception

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1998-01

PRIMARY OUTCOMES:
Disease-free survival | 24 months
Overall Survival | 24 months

SECONDARY OUTCOMES:
Immune Reconstitution | over 24 months
Organ-specific response parameters | 24 months
Serological Response (Autoantibodies) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Renate Arnold, Prof. Dr. med., Principal Investigator — Charite University, Berlin, Germany; Falk Hiepe, Prof. Dr. med., Study Chair — Charite University, Berlin, Germany
Locations (1):
- Charité Universitätsmedizin Berlin, Berlin, Germany

REFERENCES:
- [Result] Rosen O, Thiel A, Massenkeil G, Hiepe F, Haupl T, Radtke H, Burmester GR, Gromnica-Ihle E, Radbruch A, Arnold R. Autologous stem-cell transplantation in refractory autoimmune diseases after in vivo immunoablation and ex vivo depletion of mononuclear cells. Arthritis Res. 2000;2(4):327-36. doi: 10.1186/ar107. Epub 2000 Jun 8. PMID 11056673
- [Result] Jayne D, Passweg J, Marmont A, Farge D, Zhao X, Arnold R, Hiepe F, Lisukov I, Musso M, Ou-Yang J, Marsh J, Wulffraat N, Besalduch J, Bingham SJ, Emery P, Brune M, Fassas A, Faulkner L, Ferster A, Fiehn C, Fouillard L, Geromin A, Greinix H, Rabusin M, Saccardi R, Schneider P, Zintl F, Gratwohl A, Tyndall A; European Group for Blood and Marrow Transplantation; European League Against Rheumatism Registry. Autologous stem cell transplantation for systemic lupus erythematosus. Lupus. 2004;13(3):168-76. doi: 10.1191/0961203304lu525oa. PMID 15119545
- [Result] Rosen O, Hiepe F, Massenkeil G, Thiel A, Arnold R. Relapse of systemic lupus erythematosus. Lancet. 2001 Mar 10;357(9258):807-8. doi: 10.1016/S0140-6736(05)71239-3. No abstract available. PMID 11254005
- [Result] Thiel A, Alexander T, Schmidt CA, Przybylski GK, Kimmig S, Kohler S, Radtke H, Gromnica-Ihle E, Massenkeil G, Radbruch A, Arnold R, Hiepe F. Direct assessment of thymic reactivation after autologous stem cell transplantation. Acta Haematol. 2008;119(1):22-7. doi: 10.1159/000117824. Epub 2008 Feb 22. PMID 18292651
- [Result] Rosen O, Massenkeil G, Hiepe F, Pest S, Hauptmann S, Radtke H, Burmester G, Thiel A, Radbruch A, Heymer B, Arnold R. Cardiac death after autologous stem cell transplantation (ASCT) for treatment of systemic sclerosis (SSc): no evidence for cyclophosphamide-induced cardiomyopathy. Bone Marrow Transplant. 2001 Mar;27(6):657-8. doi: 10.1038/sj.bmt.1702829. PMID 11319598
- [Derived] Alexander T, Thiel A, Rosen O, Massenkeil G, Sattler A, Kohler S, Mei H, Radtke H, Gromnica-Ihle E, Burmester GR, Arnold R, Radbruch A, Hiepe F. Depletion of autoreactive immunologic memory followed by autologous hematopoietic stem cell transplantation in patients with refractory SLE induces long-term remission through de novo generation of a juvenile and tolerant immune system. Blood. 2009 Jan 1;113(1):214-23. doi: 10.1182/blood-2008-07-168286. Epub 2008 Sep 29. PMID 18824594